CLINICAL TRIAL: NCT04282538
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation as Adjunctive Rehabilitation for Cerebrovascular Disease-related Gait Dysfunction
Brief Title: Efficacy of rTMS and tDCS as Adjunctive Rehabilitation for Cerebrovascular Disease-related Gait Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: zsneurology (Other)
Responsible Party: Sponsor-Investigator, zsneurology, Medical doctor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17411953800
Record Dates: First submitted 2019-07-25; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Repetitive Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation; Cerebrovascular Disease; Gait Dysfunction, Neurologic
MeSH Terms: conditions — Cerebrovascular Disorders; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A - Active (Active Comparator): Active rTMS for Gait Dysfunction of Hemiplegia
  Interventions: Device: Active rTMS; Other: Walking training
- Group A - Sham (Sham Comparator): Sham rTMS for Gait Dysfunction of Hemiplegia
  Interventions: Device: Sham rTMS; Other: Walking training
- Group B - Active (Active Comparator): Active tDCS for Frontal Gait Dysfunction
  Interventions: Device: Active tDCS; Other: Walking training; Other: Cognition training
- Group B - Sham (Sham Comparator): Sham tDCS for Frontal Gait Dysfunction
  Interventions: Device: Sham tDCS; Other: Walking training; Other: Cognition training

INTERVENTIONS:
Device: Active rTMS — 4-week (5 days per week) active rTMS (90%rMT, M1, 10Hz for 10s, 50s interval, 20 trains)
  Arms: Group A - Active
Device: Sham rTMS — 4-week (5 days per week) sham rTMS
  Arms: Group A - Sham
Device: Active tDCS — 4-week (5 days per week) active tDCS (2mA, DLPFC, 20 min)
  Arms: Group B - Active
Device: Sham tDCS — 4-week (5 days per week) sham tDCS
  Arms: Group B - Sham
Other: Walking training — 4-week (5 days per week) walking training
Other: Cognition training — 4-week (5 days per week) cognition training
  Arms: Group B - Active; Group B - Sham

SUMMARY:
This study was a prospective, randomized, single-blind, parallel-controlled, multicenter clinical study to evaluate the efficacy and safety of repetitive transcranial magnetic stimulation and transcranial direct current stimulation assisted rehabilitation in the treatment of cerebrovascular disease-related gait disorders.

DETAILED DESCRIPTION:
This study was a prospective, randomized, single-blind, parallel-controlled, multicenter clinical study. The main purpose was to evaluate the efficacy and safety of repetitive transcranial magnetic stimulation and transcranial direct current stimulation assisted rehabilitation in the treatment of cerebrovascular disease-related gait disorders. The secondary objective was to assess the effects of these two types of neuromodulation on cognitive, emotional, and daily living abilities.

ELIGIBILITY:
Inclusion Criteria:

1. Group A: Gait Dysfunction of Hemiplegia

   * Age ≥ 35 years old, ≤ 75 years old;
   * There was a cerebral infarction event in the past ≥ 2 months, leaving unilateral lower extremity paralysis, muscle strength IV to V- grade;
   * Brunnstrom staging: lower limb of paralysis (IV-V grade), lower limb of healthy side (IV-V grade), upper limbs (IV-V grade), hands (IV-V grade);
   * Able to stand for 5 minutes without assistance, without gait aid, and to walk independently for 5 minutes without stopping;
   * Mini-mental state examination (MMSE) > 17 points, able to complete cognitive and gait assessments.
2. Group B: Frontal Gait Dysfunction

   * Age ≥ 35 years old, ≤ 75 years old;
   * Meet the frontal gait characteristics: a) Balance dysfunction: wide step base, trunk swing, increased fall, decreased trunk movement control, and autonomous activity dysfunction; b) difficulty in starting, dragging and freezing; c) without limb ataxia, dysarthria, nystagmus, decreased facial expression, decreased upper limb joint activity, upper motor neuron impaired signs, and resting tremor;
   * There was a cerebral infarction event ≥ 2 months, or asymptomatic stroke event but the head MRI suggested single or multiple lacunar infarction or ischemic lesion (diameter ≤ 2cm);
   * limb muscle strength V- to V grade, and the muscle strength of both limbs is the same;
   * Able to stand for 5 minutes without assistance, without gait aid, to walk independently for 5 minutes;
   * Able to complete cognitive and gait assessments.

Exclusion Criteria:

* Other gait abnormalities caused by other diseases, such as Parkinson's disease, hydrocephalus, cerebellar disease, vestibular system disease, extrapyramidal abnormalities, abnormalities of proprioceptive sensibility, visual abnormalities, auditory abnormalities, peripheral nerves and musculoskeletal diseases;
* Symptomatic cerebral infarction <2 months; Severe nervous system diseases, such as previous cerebral hemorrhage, history of subarachnoid hemorrhage, craniocerebral trauma, cerebral vascular malformation, brain tumor, central nervous system infection, demyelinating disease, epilepsy, myelopathy, etc.;
* Severe cognitive impairment, major depression, and aphasia disable to finish the cognitive and gait assessments;
* serious cardiovascular, pulmonary, blood, rheumatism and other complications, pregnancy;
* Metal implants such as pacemakers or cochlear implants;
* Taking drugs that affect cortical excitability: such as antiepileptic drugs, sedation, benzodiazepines, antidepressants, dopamine, amphetamines, etc.;
* long-term heavy drinking: the alcohol content of men drinking more than 168g per week, women more than 112g;
* Neurological rehabilitation treatment was received within 1 month before the start of the trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Velocity of 10m walking test | 12 weeks
  Velocity of 10m walking test (10MWT) according to the video

SECONDARY OUTCOMES:
10m walking test | 12 weeks
  Step width, step size, step frequency of 10m walking test (10MWT) according to the video
Turn time of time up and go test | 12 weeks
  Total time, pace, standing time, turn time of time up and go test (TUGT) according to the video
Dual-task walking | 12 weeks
  Pace, step width, step size, step frequency, dual task cost of dual-task walking (DTW) according to the video
Tinetti Balance and Gait Analysis | 12 weeks
  Gait evaluation according to Tinetti Balance and Gait Analysis (Full score: 28. score >= 19 indicates high risk of fall.)
Mini-mental state examination (MMSE) | 12 weeks
  Cognition evaluation according to Mini-mental state examination (Full score: 30. score <24 indicates cognitive impairment. )
Montreal cognitive assessment (MoCA) | 12 weeks
  Cognition evaluation according to Montreal cognitive assessment (Full score: 30. score <26 indicates cognitive impairment.
Symbol digit modalities test (SDMT) | 12 weeks
  Attention evaluation according to Symbol digit modalities test (Counting number of right modalities in 90s. )
Color word test (CWT) | 12 weeks
  Execution evaluation according to Color word test (Counting number of right ones. )
Hamilton depression scale (HAMD) | 12 weeks
  Mood evaluation according to Hamilton depression scale (Score >7 indicates possible depression.)
Instrumental activities of daily living (IADL) | 12 weeks
  Daily living ability evaluation according to Instrumental activities of daily living (Full score: 24. Higher score indicates higher independence. )

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (6):
- China (6):
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Eighth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Huadong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No